CLINICAL TRIAL: NCT07356622
Title: The Assessment of The Volumetric Occlusal Adjustments Required for Michigan Splints Fabricated Using Various Digital Bite Registrations
Brief Title: Occlusal Adjustments Needed for Michigan Splints Made Using Different Digital Bite Records
Acronym: AVOAMSDBR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Guy's Hospital (Other)
Responsible Party: Principal Investigator, Arwa Alhusban, Dr Arwa Ibrahim Alhusban, King's College London
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 43439; HR2301469 (Other Grant/Funding Number: The Hashemite university of Jordan)
Record Dates: First submitted 2026-01-05; First posted 2026-01-21 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Temporomandibular Disorders (TMD)
Keywords: Digital occlusal recording; Digital bite registration; Occlusal splint fabrication; Occlusal splint accuracy; Michigan splint; Digital facebow; Virtual articulator; Three-dimensional printing
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Intervention Model Description: Participants undergo multiple digital bite registration procedures. Michigan occlusal splints fabricated using each method are assessed within the same participant, allowing within-subject comparison of occlusal accuracy and root mean square (RMS) deviation.
Who Masked: Participant
Masking Description: Participants are blinded to the type of digital bite registration method used to fabricate each of the four Michigan occlusal splints. Each participant is required to try four splints in a crossover manner, with splints coded and presented in identical appearance so that participants cannot distinguish which recording method was used for any given splint. Clinicians and researchers involved in splint fabrication and assessment are not blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Retruded axis position(RAP with) without a digital facebow (Experimental): Each participant received Michigan occlusal splints fabricated using digital bite registration methods, including Retruded axis position(RAP with) without a digital facebow. Participants try each splint in a crossover manner while being blinded to the recording method used. Occlusal accuracy and adjustment requirements are evaluated using three-dimensional surface superimposition and root mean square (RMS) deviation analysis.
  Interventions: Device: Digital face-bow, digital bite registration, digital scanning
- Retruded axis position(RAP) with a digital facebow. (Experimental): Each participant received Michigan occlusal splints fabricated using digital bite registration methods, including Retruded axis position(RAP) with a digital facebow. Participants try each splint in a crossover manner while being blinded to the recording method used. Occlusal accuracy and adjustment requirements are evaluated using three-dimensional surface superimposition and root mean square (RMS) deviation analysis.
  Interventions: Device: Digital facebow, digital bite registration, digital scanning
- Intercuspal position (ICP) with a digital facebow (Experimental): Each participant received Michigan occlusal splints fabricated using digital bite registration methods, including maximum intercuspal position (ICP) with a digital facebow. Participants try each splint in a crossover manner while being blinded to the recording method used. Occlusal accuracy and adjustment requirements are evaluated using three-dimensional surface superimposition and root mean square (RMS) deviation analysis.
  Interventions: Device: Retruded axis position(RAP with) without a digital facebow
- Intercuspal position (ICP) without a digital facebow. (Experimental): Each participant received Michigan occlusal splints fabricated using digital bite registration methods, including maximum intercuspal position (ICP) without a digital facebow. Participants try each splint in a crossover manner while being blinded to the recording method used. Occlusal accuracy and adjustment requirements are evaluated using three-dimensional surface superimposition and root mean square (RMS) deviation analysis.
  Interventions: Device: Digital face-bow, digital bite registration, digital scanning

INTERVENTIONS:
Device: Retruded axis position(RAP with) without a digital facebow — The intervention involves the fabrication of Michigan occlusal splints using different digital bite registration workflows. Each participant undergoes digital occlusal recording in centric relation (CR) and intercuspal position (ICP), with and without the use of an Axioprisa® digital facebow, and articulation is performed using Axioprisa® virtual articulator. Four splints are fabricated per participant based on these recordings. Participants are blinded to the recording method used for each splint and try all splints in a crossover manner. Occlusal accuracy and adjustment requirements are evaluated using three-dimensional surface superimposition and root mean square (RMS) deviation analysis.
  Arms: Intercuspal position (ICP) with a digital facebow
Device: Digital face-bow, digital bite registration, digital scanning — The intervention involves the fabrication of Michigan occlusal splints using different digital bite registration workflows. Each participant undergoes digital occlusal recording in centric relation (CR) and intercuspal position (ICP), with and without the use of an Axioprisa® digital facebow, and articulation is performed using Axioprisa® virtual articulator. Four splints are fabricated per participant based on these recordings. Participants are blinded to the recording method used for each splint and try all splints in a crossover manner. Occlusal accuracy and adjustment requirements are evaluated using three-dimensional surface superimposition and root mean square (RMS) deviation analysis.
  Arms: Intercuspal position (ICP) without a digital facebow.; Retruded axis position(RAP with) without a digital facebow
Device: Digital facebow, digital bite registration, digital scanning — The intervention involves the fabrication of Michigan occlusal splints using different digital bite registration workflows. Each participant undergoes digital occlusal recording in centric relation (CR) and intercuspal position (ICP), with and without the use of an Axioprisa® digital facebow, and articulation is performed using Axioprisa® virtual articulator. Four splints are fabricated per participant based on these recordings. Participants are blinded to the recording method used for each splint and try all splints in a crossover manner. Occlusal accuracy and adjustment requirements are evaluated using three-dimensional surface superimposition and root mean square (RMS) deviation analysis.
  Arms: Retruded axis position(RAP) with a digital facebow.

SUMMARY:
This clinical study evaluated digital occlusal recording methods used in the fabrication of Michigan occlusal splints. The objective was to assess whether different digital bite registration techniques influenced the accuracy of occlusal splints and the amount of occlusal adjustment required at clinical fitting.

Participants underwent digital bite registration procedures and received Michigan occlusal splints fabricated using different digital workflows. Follow-up visits were conducted for splint fitting and occlusal assessment. Participant safety and data confidentiality were maintained throughout the study, and all required ethical approvals and risk assessments were obtained prior to study initiation.

The study findings were intended to support improvements in digital dental workflows and enhance the accuracy and efficiency of occlusal splint fabrication.

DETAILED DESCRIPTION:
Background Temporomandibular disorders represented a common clinical condition affecting mandibular function and were frequently associated with parafunctional activities such as bruxism or clenching. Clinical features included orofacial pain, joint sounds, restricted mandibular movement, headaches, dental wear, and occlusal instability. Occlusal splints were commonly prescribed to reduce occlusal loading, protect dental structures, and establish a more favourable mandibular position.

Conventional occlusal splint fabrication relied on physical impressions, mechanical articulation, and manual occlusal adjustment. These processes were time-consuming and technique-sensitive. Digital dentistry introduced alternative workflows incorporating intraoral scanning, virtual articulation, and computer-aided design and manufacturing, with the aim of improving accuracy, reproducibility, and efficiency.

Accurate digital recording of the maxillomandibular relationship remained a critical factor influencing occlusal outcomes. Digital bite registration techniques performed at intercuspal position or centric relation, with or without digital facebow transfer, were expected to affect occlusal accuracy and the extent of chairside adjustment required at delivery.

Virtual articulators were developed to simulate mandibular movements using digitally acquired data. These systems required accurate digital impressions, occlusal records, and appropriate orientation of the maxillary arch relative to craniofacial reference planes. Digital facebow systems enabled virtual transfer of maxillary position and were expected to improve mounting accuracy compared with average-value articulators alone.

Study objectives Primary Objectives

* To evaluate volumetric changes on the occlusal surfaces of Michigan splints following clinical adjustment.
* To compare pre-adjustment and post-adjustment occlusal surface volumes across different digital workflows.
* To assess whether an average-value virtual articulator produced occlusal splints at an increased occlusal vertical dimension without the need for clinical registration.

Secondary objectives

* To assess laboratory efficiency and quality control associated with digital workflows.
* To evaluate clinical time and effort required for occlusal adjustment.
* To assess participant comfort during digital recording procedures.

This was a single-centre clinical study involving 10 participants. Each participant received four Michigan occlusal splints, corresponding to four different digital design workflows based on mandibular recording position and the inclusion or exclusion of a digital facebow record. Each of the four digital designs generated for every participant was manufactured as a separate occlusal splint, resulting in four splints per participant.

Clinical and laboratory procedures Visit 1

* Informed consent was obtained.
* Standardised dental photography was performed.
* A digital facebow record was obtained using a digital facebow system equipped with a scannable bite fork (Axiopresia) as part of the registration process, where applicable. The scannable bite fork was positioned intraorally and digitally captured to record the spatial relationship of the maxillary arch relative to craniofacial reference planes.
* Digital impressions of the maxillary and mandibular arches were obtained using an intraoral scanner under standardised clinical conditions.
* Bite registration at centric relation/ retruded articulation position was obtained following neuromuscular deprogramming using a Lucia gauge and intraoral scanner.
* Bite registration at intercuspal position was recorded using the intraoral scanner.

Laboratory procedures

Using computer-aided design software, four distinct digital occlusal splint designs were produced for each participant based on different combinations of mandibular recording position and digital facebow transfer:

Retruded articulation position (centric relation) with digital facebow record Retruded articulation position (centric relation) without digital facebow record Intercuspal position with digital facebow record Intercuspal position without digital facebow record Each digital design was generated using the same virtual articulator parameters and identical splint design settings, differing only in the mandibular position record and the inclusion or exclusion of the digital facebow data. The resulting designs were then manufactured using three-dimensional printing.

Visit 2: Fitting and occlusal adjustment

* Clinical fitting of the occlusal splints was performed during the second visit.
* Occlusal adjustments were carried out to achieve balanced light occlusal contacts at the resting intercuspal position.
* Lateral movements were assessed to confirm canine guidance, and anterior guidance was evaluated during protrusive movements.
* Any occlusal interferences were identified and removed accordingly to achieve a stable and harmonious occlusal scheme.
* Following completion of occlusal adjustments, the splints were digitally scanned via lab scanner for post-adjustment analysis.

Outcome assessment Pre-adjustment and post-adjustment digital scans of each occlusal splint were imported into three-dimensional analysis software ( Geomagic software). Root mean square deviation values were calculated following best-fit alignment to quantify volumetric changes associated with occlusal adjustment. The 3D and 2D Comparisons at six sections were done ( middle of the cingulum of the right and left central incisor, middle of the cingulum of the right and left canines, messy-buccal cusp to disco-palatal cup of the right and left first molar). Occlusal deviation maps were standardised using consistent colour scales to allow comparison between workflows.

ELIGIBILITY:
Inclusion Criteria:•

* Aged between 18 and 65.
* Able to provide informed consent.
* Have no more than one tooth missing per quadrant.

Exclusion Criteria:

* Patients with removable dentures
* Patients receiving medication for psychological disorders.
* Patients diagnosed with systemic joint disorders.
* Pregnant.
* Patients who have received TMD treatment in the last 6 months.
* Deep bite cases.
* Those who have an extreme class 3 dental or skeletal relationship.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Volumetric occlusal adjustment of michigan occlusal splints | Baseline (pre-adjustment) and at splint fitting (post-adjustment)
  The primary outcome was the volume of occlusal adjustment required for Michigan occlusal splints fabricated using different digital bite registration workflows. Volumetric changes were quantified by calculating root mean square (RMS) deviation values between pre-adjustment and post-adjustment digital scans of each splint using three-dimensional surface comparison software. Higher RMS values indicated greater occlusal adjustment.

SECONDARY OUTCOMES:
Occlusal contact quality after adjustment of michigan occlusal splints | At splint fitting visit
  The secondary outcome was the qualitative assessment of occlusal contact quality following clinical adjustment of Michigan occlusal splints fabricated using different digital workflows. Occlusion was assessed clinically to confirm balanced light contacts at the resting intercuspal position, presence of canine guidance during lateral excursions, presence of anterior guidance during protrusive movements, and elimination of occlusal interferences. Outcomes were recorded as achievement of a stable and clinically acceptable occlusal scheme following adjustment.

OTHER OUTCOMES:
Pattern of occlusal adjustment on splints after fitting | Baseline (before adjustment) and at splint fitting
  This outcome examined where occlusal adjustments occurred on Michigan occlusal splints after clinical fitting. Digital scans of each splint taken before and after adjustment were compared using computer software to show areas where material was removed. The comparison included both an overall surface assessment and simple two-dimensional comparisons at the front (anterior) and back (posterior) areas of the splint. This helped describe how occlusal adjustments were distributed across different parts of the splint for each digital design.

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, Sothwarck, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the small sample size and the potentially identifiable nature of dental imaging and 3D surface data. Aggregate, anonymised results will be reported.

REFERENCES:
- [Background] Obrez A, et al. Accuracy of opening the vertical dimension on virtual articulators. J Prosthodont. 2019.
- [Background] 1-Gross MD. The facebow: Use, misuse, and abuse. J Prosthet Dent. 1982;48:377-382.
- See also: Clinical trial ethics websute — https://internal.kcl.ac.uk/innovation/clinical-trials/index

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2024-07-23): https://cdn.clinicaltrials.gov/large-docs/22/NCT07356622/Prot_SAP_000.pdf
  • Informed Consent Form: patient information sheet (2024-07-13): https://cdn.clinicaltrials.gov/large-docs/22/NCT07356622/ICF_001.pdf
  • Informed Consent Form: Informed consent formt (2024-07-13): https://cdn.clinicaltrials.gov/large-docs/22/NCT07356622/ICF_002.pdf